CLINICAL TRIAL: NCT00831857
Title: 89Zr-bevacizumab PET Imaging in Patients With Renal Cell Carcinoma Treated With Sunitinib or Bevacizumab Plus Interferon; a Pilot Study
Brief Title: VEGF Imaging in Renal Cell Carcinoma
Acronym: Renimage
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: Renimage Protocol
Record Dates: First submitted 2009-01-28; First posted 2009-01-29 (Estimated); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A: Treatment with sunitinib.
  Interventions: Other: 89Zr-Bevacizumab PET-scan
- Group B: Treatment with bevacizumab and interferon
  Interventions: Other: 89Zr-Bevacizumab PET-scan

INTERVENTIONS:
Other: 89Zr-Bevacizumab PET-scan — At baseline, after two weeks of treatment and after 6 weeks of treatment.

SUMMARY:
The primary objective of the study is to evaluate the feasibility of 89Zr-bevacizumab PET imaging as a biomarker before and during treatment with sunitinib or bevacizumab plus interferon in patients with RCC. 89Zr-bevacizumab PET imaging will be regarded a promising biomarker if the target for treatment (VEGF) can be visualised and if uptake changes after institution of treatment.

DETAILED DESCRIPTION:
* To explore if 89Zr-bevacizumab PET imaging can differentiate RCC patients with progressive disease from patients with non-progressive disease during treatment with sunitinib or bevacizumab plus interferon.
* To explore relationships between VEGF pathway related biomarkers and 89Zr-bevacizumab PET response.
* To explore effect of 2 weeks off treatment in the sunitinib arm on pharmacodynamic biomarkers and 89Zr-bevacizumab PET response.

ELIGIBILITY:
Inclusion criteria:

* locally advanced irresectable or metastatic renal cell cancer
* no untreated brain metastases (CT or MRI not necessary in the absence of symptoms)
* no uncontrolled hypertension
* no clinically significant cardiovascular events or disease during the last 12 months
* no surgery in the last 4 weeks
* no treatment with bevacizumab or another monoclonal antibody with anti-angiogenic properties in the last 4 months
* no treatment with a tyrosine kinase inhibitor during the last 4 weeks
* measurable disease with x-ray or CT scan, at least one site of disease must be unidimensionally measurable as follows: X-ray > 20 mm, Spiral CT scan > 10 mm, non-spiral CT scan > 20 mm
* clear cell histology component
* not pregnant or nursing
* women of childbearing potential must use effective contraception
* absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* before patient randomization, written informed consent must be given according to GCP, and local regulations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients locally advanced irresectable or metastatic renal cell cancer.
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2009-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the change in SUV between baseline 89Zr-bevacizumab PET scan and the scan performed after 2 and 6 weeks of treatment with sunitinib or bevacizumab plus interferon in patients with RCC. | after 2 and 6 weeks

SECONDARY OUTCOMES:
Progressive disease according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria. Progression is defined as the appearance of new disease or an increase of 20% in the sum of the longest diameters of the target lesions. | 3 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sjoukje F. Oosting, MD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands